CLINICAL TRIAL: NCT06428942
Title: Increased Low-potassium Content Vegetables Consumption in Patients With Moderate-to-severe Chronic Kidney Disease: a Randomized Controlled Trial
Brief Title: Low-potassium Content Vegetables in Chronic Kidney Disease
Acronym: LPV in CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Szu-Chun Hung, Professor, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-XD-093
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: the Recommended Target of Daily Vegetables Intake; Risk of Hyperkalemia
Keywords: chronic kidney disease; vegetables; hyperkalemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia

STUDY DESIGN:
Intervention Model Description: Participants are randomized to intervention group or control group with ratio of 50:25.
Masking Description: Masking is not allowed in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants in the intervention group would receive their daily low-potassium vegetables 3 to 5 serving according to their daily suggested requirement and routine CKD dietary education for 8 weeks.
  Interventions: Other: low-potassium vegetables
- Control group (No Intervention): The participants in the control group would receive routine CKD dietary education for 8 weeks.

INTERVENTIONS:
Other: low-potassium vegetables — low-potassium vegetables 3 to 5 serving according to their daily suggested requirement
  Arms: Intervention group

SUMMARY:
Prior observational studies have shown that higher levels of vegetables and fruits consumption are associated with lower risk of all-cause mortality in patients with chronic kidney disease (CKD). However, compared with the normal population, patients with CKD are more likely to consume less vegetables and fruits. Thus, the investigators aim to evaluate whether proving low-potassium content vegetables to this population are able to reach the recommended target of daily vegetables intake and not increase the risk of hyperkalemia.

DETAILED DESCRIPTION:
Prior observational studies have shown that higher levels of vegetables and fruits consumption are associated with lower risk of all-cause mortality in patients with chronic kidney disease (CKD). However, compared with the normal population, patients with CKD are more likely to consume less vegetables and fruits. According to the suggestions from 2018 Ministry of Health and Welfare in Taiwan, vegetables intake are at least 3 to 5 servings daily based on the daily energy requirement. In our own data, the average daily vegetables intake was only 2.1 servings among patients with CKD stages 3 to 5 not yet on dialysis. Therefore, the investigators aim to evaluate whether proving low-potassium content vegetables to patients with CKD stages 3 to 5 not yet on dialysis are able to reach the recommended target of daily vegetables intake and not increase the risk of hyperkalemia.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 3b~5, not yet on dialysis
* Age ≥20 years
* Stable doses of medications for 4 weeks
* Serum potassium level: ≥3.5 and < 5.5 mmol/L

Exclusion Criteria:

* Anticipated to receive dialysis within 3 month
* Major gastrointestinal diseases (inflammatory bowel disease, celiac disease) or intestinal resection
* Patients with infection, malignancy, heart failure, liver cirrhosis or impaired cognitive or mental disorders
* Patients who are just hospitalized due to an acute cardiovascular events or infection 3 months prior to the start of study
* Patients with kidney transplants
* Patients who receive immunosuppressant
* Pregnant women or patients who are planning to become pregnant

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-05-27 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who reach the targets of daily vegetable recommended target | 8 weeks
  Percentage of participants who reach the targets of daily vegetable recommended

SECONDARY OUTCOMES:
Gut-derived uremic toxins | 8 weeks
  Change in gut-derived uremic toxins ( indoxyl sulfate, p-cresyl sulfate)
Serum creatinine | 8 weeks
  Change in serum creatinine in mg/dL
Proteinuria | 8 weeks
  Change in proteinuria in g/day
Occurrence of moderate hyperkalemia | 8 weeks
  serum [potassium] >=5.5 mmol/L
Status of constipation | 8 weeks
  Using the Chinese constipation questionnaire. The minimum value is 0, and the maximum value is 21, and the higher score represents a worse outcome.
Gut microbiome | 8 weeks
  Change in alpha- and beta-diversities indices

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Chun Hung, MD, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
We do not have IPD sharing plan.

REFERENCES:
- [Background] Wakasugi M, Yokoseki A, Wada M, Momotsu T, Sato K, Kawashima H, Nakamura K, Onodera O, Narita I. Vegetable and Fruit Intake Frequency and Mortality in Patients With and Without Chronic Kidney Disease: A Hospital-Based Cohort Study. J Ren Nutr. 2023 Jul;33(4):566-574. doi: 10.1053/j.jrn.2023.01.011. Epub 2023 Feb 13. PMID 36791982
- [Background] Saglimbene VM, Wong G, Ruospo M, Palmer SC, Garcia-Larsen V, Natale P, Teixeira-Pinto A, Campbell KL, Carrero JJ, Stenvinkel P, Gargano L, Murgo AM, Johnson DW, Tonelli M, Gelfman R, Celia E, Ecder T, Bernat AG, Del Castillo D, Timofte D, Torok M, Bednarek-Skublewska A, Dulawa J, Stroumza P, Hoischen S, Hansis M, Fabricius E, Felaco P, Wollheim C, Hegbrant J, Craig JC, Strippoli GFM. Fruit and Vegetable Intake and Mortality in Adults undergoing Maintenance Hemodialysis. Clin J Am Soc Nephrol. 2019 Feb 7;14(2):250-260. doi: 10.2215/CJN.08580718. Epub 2019 Jan 31. PMID 31738182
- [Background] Pourafshar S, Sharma B, Kranz S, Mallawaarachchi I, Kurland E, Ma JZ, Scialla JJ. Patterns of Fruit and Vegetable Intake in Adults With and Without Chronic Kidney Disease in the United States. J Ren Nutr. 2023 Jan;33(1):88-96. doi: 10.1053/j.jrn.2022.06.007. Epub 2022 Jul 5. PMID 35798188